CLINICAL TRIAL: NCT06751654
Title: Can Total Mechanical Power Be a Determinant of Weaning Failure in Chronic Obstructive Pulmonary Disease (COPD)?
Status: Completed | Type: Observational
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Collaborators: Masih Daneshvari Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-12-06
Record Dates: First submitted 2024-12-11; First posted 2024-12-30 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease); ARDS (Acute Respiratory Distress Syndrome); Mechanical Power; Pneumonia; Weaning Failure
Keywords: Mechanical Power; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Acute Lung Injury; Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Weaned: patients with successful weaning from mechanic ventilator
- Non-weaned: patients who have failed to wean from ventilator

SUMMARY:
A Comparison of Ventilator Parameters (TV, DP, Total Mechanical Power, etc.) Between Successfully and unsuccessfully Weaned Patients with COPD Undergoing Mechanical Ventilation Due to Respiratory Failure, and Diagnosed with Pneumonia or ARDS in the Intensive Care Unit."

DETAILED DESCRIPTION:
The objective of this study is to investigate which mechanical ventilation parameters and clinical findings influence weaning success by comparing successful and unsuccessful weaning patient groups among patients diagnosed with COPD who were intubated and monitored for more than five days in the intensive care unit. The findings of this study may contribute to the development of future treatment protocols and criteria for evaluating the weaning process.

This study is planned to be conducted in two centers: Bakırköy Dr. Sadi Konuk Training and Research Hospital in Istanbul and Shahid Beheshti University of Medical Sciences, Masih Daneshvari Hospital in Tehran. This multicenter study aims to facilitate the comparison of data obtained under different geographical and clinical conditions, thereby enabling a broader analysis of factors influencing the weaning process across a larger patient population.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older
* COPD-diagnosed patients who have been intubated and stayed in the ICU for more than 5 days

Exclusion Criteria:

* Patients without electronic medical records
* Patients under 18 years of age
* Patients diagnosed with pulmonary malignancy
* Patients who stayed in the ICU for less than 5 days
* Patients monitored in the ICU without intubation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intubated patients with COPD which has been diagnosed Pneumonia or ARDS and have admission to icu and stayed for more than 5 years.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2024-12-06 (Actual); Primary Completion 2024-12-23 (Actual); Study Completion 2024-12-23 (Actual)

PRIMARY OUTCOMES:
Successful Weaning | 48 hours
  The primary outcome of this study will be the successful weaning from mechanical ventilation. This will be defined as the patient being successfully extubated and maintaining adequate oxygenation for more than 48 hours without requiring reintubation or mechanical ventilation support.

SECONDARY OUTCOMES:
Mechanical Ventilator Parameters | 48 hours
  A comparison of total mechanical power between the weaned and non-weaned patient groups.

CONTACTS AND LOCATIONS:
Overall Officials: Zafer Cukurova, M.D, Study Chair — Bakırkoy Dr. Sadi Konuk Training and Research Hospital; Seyed Mohammadreza Hashemian, M.D, Study Director — Masih Daneshvari Hospital
Locations (1):
- Bakirkoy Dr Sadi Konuk Research and Training Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No